CLINICAL TRIAL: NCT06096077
Title: Evaluation of Tranexamic Acid for Angiotensin-converting Enzyme Inhibitor-induced Angioedema in the Emergency Department
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 114.PHA.2022.C
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Angioedema
MeSH Terms: conditions — Angioedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective Cohort: ED at MCMC for ACEi-AE with TXA
- Retrospective Chort: ED at MCMC for ACEi-AE without TXA

SUMMARY:
Angiotensin-converting enzyme inhibitor ACEi induced angioedema ACEi-AE is defined as physical swelling of the deep skin layers or mucous membranes due to increased vascular permeability and leakage of fluid into the interstitial space caused while taking an ACEi

DETAILED DESCRIPTION:
Angiotensin-converting enzyme inhibitor ACEi induced angioedema ACEi-AE most commonly affects the lips, mouth, face, upper airway, and less commonly the gastrointestinal tract. This condition may lead to life-threatening airway compromise which would require emergent intubation. Currently, strong evidence is lacking to help guide management of ACEi-AE in the emergency department (ED).

ELIGIBILITY:
Inclusion Criteria:

•Patients must be ≥ 18 years old, be diagnosed with suspected ACEi-AE (with ACEi use). ACEi use is defined as patient-reported use or evidence indicating use listed in the chart.

Exclusion Criteria:

•Patients will be excluded if they have an allergy to TXA or any components of the formulation, present with an urticaria, have a personal or family history of hereditary angioedema, or received TXA administration in another department besides the ED.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must be ≥ 18 years old, be diagnosed with suspected ACEi-AE (with ACEi use). ACEi use is defined as patient-reported use or evidence indicating
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-08-23 (Actual)

PRIMARY OUTCOMES:
Intubation patients | 2 weeks
  Proportion of patients who required intubation during their hospital length of stay.
Admission proportion | 2 weeks
  The proportion of admissions to the ICU or another floor within MCMC Time to hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Lin, PharmD, Principal Investigator — Methodist Charlton Medical Center
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Study data or any protected health information will not be shared with anyone that is not delegated to the study. The PI is committed to disseminate research results in a timely fashion. Sharing of results generated by the data analysis during the course of the project will be through presentation at national scientific meetings and/or publication in open access journals. All information obtained will be source de-identified and presented on a large scale and not traceable to any one particular individual.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 2 years

REFERENCES:
- [Background] Moellman JJ, Bernstein JA, Lindsell C, Banerji A, Busse PJ, Camargo CA Jr, Collins SP, Craig TJ, Lumry WR, Nowak R, Pines JM, Raja AS, Riedl M, Ward MJ, Zuraw BL, Diercks D, Hiestand B, Campbell RL, Schneider S, Sinert R; American College of Allergy, Asthma & Immunology (ACAAI); Society for Academic Emergency Medicine (SAEM). A consensus parameter for the evaluation and management of angioedema in the emergency department. Acad Emerg Med. 2014 Apr;21(4):469-84. doi: 10.1111/acem.12341. PMID 24730413
- [Background] Zuraw BL, Bernstein JA, Lang DM, Craig T, Dreyfus D, Hsieh F, Khan D, Sheikh J, Weldon D, Bernstein DI, Blessing-Moore J, Cox L, Nicklas RA, Oppenheimer J, Portnoy JM, Randolph CR, Schuller DE, Spector SL, Tilles SA, Wallace D; American Academy of Allergy, Asthma and Immunology; American College of Allergy, Asthma and Immunology. A focused parameter update: hereditary angioedema, acquired C1 inhibitor deficiency, and angiotensin-converting enzyme inhibitor-associated angioedema. J Allergy Clin Immunol. 2013 Jun;131(6):1491-3. doi: 10.1016/j.jaci.2013.03.034. PMID 23726531
- [Background] Banerji A, Clark S, Blanda M, LoVecchio F, Snyder B, Camargo CA Jr. Multicenter study of patients with angiotensin-converting enzyme inhibitor-induced angioedema who present to the emergency department. Ann Allergy Asthma Immunol. 2008 Apr;100(4):327-32. doi: 10.1016/S1081-1206(10)60594-7. PMID 18450117
- [Background] Gabb GM, Ryan P, Wing LM, Hutchinson KA. Epidemiological study of angioedema and ACE inhibitors. Aust N Z J Med. 1996 Dec;26(6):777-82. doi: 10.1111/j.1445-5994.1996.tb00624.x. PMID 9028507
- [Background] Sarkar P, Nicholson G, Hall G. Brief review: angiotensin converting enzyme inhibitors and angioedema: anesthetic implications. Can J Anaesth. 2006 Oct;53(10):994-1003. doi: 10.1007/BF03022528. PMID 16987854
- [Background] Zuraw BL. Clinical practice. Hereditary angioedema. N Engl J Med. 2008 Sep 4;359(10):1027-36. doi: 10.1056/NEJMcp0803977. No abstract available. PMID 18768946
- [Background] van den Elzen M, Go MFCL, Knulst AC, Blankestijn MA, van Os-Medendorp H, Otten HG. Efficacy of Treatment of Non-hereditary Angioedema. Clin Rev Allergy Immunol. 2018 Jun;54(3):412-431. doi: 10.1007/s12016-016-8585-0. PMID 27672078
- [Background] Bas M, Greve J, Stelter K, Havel M, Strassen U, Rotter N, Veit J, Schossow B, Hapfelmeier A, Kehl V, Kojda G, Hoffmann TK. A randomized trial of icatibant in ACE-inhibitor-induced angioedema. N Engl J Med. 2015 Jan 29;372(5):418-25. doi: 10.1056/NEJMoa1312524. PMID 25629740
- [Background] Culley CM, DiBridge JN, Wilson GL Jr. Off-Label Use of Agents for Management of Serious or Life-threatening Angiotensin Converting Enzyme Inhibitor-Induced Angioedema. Ann Pharmacother. 2016 Jan;50(1):47-59. doi: 10.1177/1060028015607037. Epub 2015 Sep 28. PMID 26416949
- [Background] Kerrigan MJ, Naik P. C1 Esterase Inhibitor Deficiency(Archived). 2023 Jul 10. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK538166/ PMID 30844193
- [Background] Busse PJ, Christiansen SC, Riedl MA, Banerji A, Bernstein JA, Castaldo AJ, Craig T, Davis-Lorton M, Frank MM, Li HH, Lumry WR, Zuraw BL. US HAEA Medical Advisory Board 2020 Guidelines for the Management of Hereditary Angioedema. J Allergy Clin Immunol Pract. 2021 Jan;9(1):132-150.e3. doi: 10.1016/j.jaip.2020.08.046. Epub 2020 Sep 6. PMID 32898710